CLINICAL TRIAL: NCT00317798
Title: A Pilot, Phase-I Trial of Rabbit Anti-Thymocyte Globulin (rATG, Thymoglobulin™) in Combination With Rapamycin in Relapsed Multiple Myeloma (MM)
Brief Title: Antithymocyte Globulin and Sirolimus in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, JJ Ifthikharuddin, Principal Investigator, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000480087; URCC-U11405; GENZ-URCC-U11405
Record Dates: First submitted 2006-04-24; First posted 2006-04-25 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: drug/agent toxicity by tissue/organ; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Antilymphocyte Serum; Sirolimus

INTERVENTIONS:
Biological: anti-thymocyte globulin — Escalating doses of rATG,intravenously, starting at 6 mg/kg to a maximum of 14.5 mg/kg. Rapamycin is given orally, starting at a dose of 1 mg daily beginning on day 1 and terminating on day 30. The dose of rapamycin was adjusted to maintain a constant blood level of 4-6 ng/ml in all subjects
Drug: sirolimus — escalating doses of rATG, intravenously, starting at 6 mg/kg to a maximum of 14.5 mg/kg. Rapamycin is given orally, starting at a dose of 1 mg daily beginning on day 1 and terminating on day 30. The dose of rapamycin was adjusted to maintain a constant blood level of 4-6 ng/ml in all subjects

SUMMARY:
RATIONALE: Biological therapies, such as antithymocyte globulin may stimulate the immune system in different ways and stop cancer cells from growing. Sirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It may also prevent or reduce the side effects of antithymocyte globulin. Giving antithymocyte globulin together with sirolimus may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of antithymocyte globulin when given together with sirolimus in treating patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability, in terms of clinical and laboratory toxicity, of anti-thymocyte globulin (ATG) combined with sirolimus in patients with relapsed multiple myeloma.
* Determine the dose-limiting toxicity of this regimen in these patients.
* Determine the maximum tolerated dose of ATG when administered with sirolimus in these patients.

Secondary

* Determine the clinical activity of this regimen, in terms of measurability of improvement in clinical benefits, in these patients.
* Assess patients for sensitivity of CD 138^-positive myeloma cells to ATG prior to treatment.
* Determine the pharmacokinetics, in terms of ATG levels in blood and bone marrow, in these patients.
* Assess the binding capability of ATG to bone marrow resident myeloma cells.
* Determine if an ATG-resistant clone emerges after treatment.

OUTLINE: This is an open-label, pilot, dose-escalation study of anti-thymocyte globulin (ATG).

Patients receive ATG IV over 6-12 hours for 4, 6, or 8 days and oral sirolimus once daily on days 1-30 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ATG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Bone marrow aspirates and blood samples are collected at baseline and periodically during study treatment for drug sensitivity and pharmacokinetic studies.

After completion of study treatment, patients are followed every 3 weeks for up to 2 months and then monthly thereafter.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously diagnosed multiple myeloma (MM) based on standard criteria

  * Soft tissue (not bone only) plasmacytomas allowed
* Measurable disease, meeting both of the following criteria:

  * Monoclonal population of plasma cell in the bone marrow
  * Quantifiable serum and/or urine monoclonal protein (i.e., generally, but not exclusively, IgG > 1 g/dL, IgA > 0.5 g/dL, or urine light-chain excretion ≥ 200 mg/24 hours)
* Steroid-refractory disease, defined as less than a minimum response to prior high-dose glucocorticoid therapy

  * Minimal response requires all of the following criteria:

    * 25-49% reduction in the level of serum monoclonal paraprotein maintained for ≥ 6 weeks
    * 50-89% reduction in 24-hour urinary light-chain excretion, but still > 200 mg/24 hours, maintained for ≥ 6 weeks
    * 25-49% reduction in the size of soft tissue plasmacytomas (clinically or by CT scan or MRI)
    * No increase in size or number of lytic bone lesions
  * High-dose glucocorticoid therapy defined as 480 mg dexamethasone (or equivalent) alone or as part of a vincristine, doxorubicin, and dexamethasone regimen
* Must have undergone autologous transplantation OR received ≥ 2 conventional lines of therapy
* Currently requiring therapy for progressive disease, as indicated by any of the following criteria:

  * 25% increase in paraprotein
  * Development of new or progression of pre-existing lytic bone lesions or soft tissue plasmacytomas
  * Hypercalcemia not attributable to any other cause
  * Relapse from complete remission
* No nonsecretory MM

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-2

  * 3-4 allowed if, in the opinion of the investigator, secondary to MM-related bone pain
* Life expectancy ≥ 3 months
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Calcium < 14 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* Hepatitis B surface antigen and hepatitis C antibody negative
* No known history of allergy to rabbit proteins
* No history of cardiac amyloidosis
* No poorly controlled hypertension, diabetes mellitus, coronary artery disease, or other serious medical or psychiatric illness
* No myocardial infarction within the past 6 weeks
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No evidence of acute ischemia or active conduction system abnormality by electrocardiogram
* No active systemic infection requiring treatment unless adequately controlled with appropriate antimicrobial therapy (e.g., treated central line infection)
* No acute viral illness
* No pathologic fractures or symptomatic hyperviscosity
* No other prior malignancy except adequately treated basal cell or squamous cell skin cancer, cervical cancer in situ, or any other cancer with a disease-free status for ≥ 3 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 8 weeks since prior immunotherapy or antibody therapy
* At least 4 weeks since prior major surgery (except for kyphoplasty)
* At least 3 weeks since prior conventional chemotherapy or radiotherapy for MM
* At least 3 weeks since prior bortezomib, thalidomide, or clarithromycin for MM
* No prior anti-thymocyte globulin
* No concurrent radiotherapy
* No other concurrent antineoplastic therapy with known activity against MM, including clarithromycin
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose | Duration of the study

SECONDARY OUTCOMES:
Relapse rates as measured by standard response criteria | Duration of the study
Laboratory correlative studies | During treatment

CONTACTS AND LOCATIONS:
Overall Officials: J. J. Ifthikharuddin, MD, Principal Investigator — James P. Wilmot Cancer Center; Martin S. Zand, MD, PhD, Principal Investigator — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States